CLINICAL TRIAL: NCT06382103
Title: Biomarkers and Molecular Mechanism Study of Hepatocellular Carcinoma After Radical Resection and Conversion Therapy
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2024-108R
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: ctDNA monitoring — The ctDNA level will be measured using tumor-informed (Signatera platform) and tumor-naived (fragmentomes measurement) assay.
Diagnostic Test: Plasma proteomic analysis — plasma protein level will be measured via Proximity Extension Assay and LC-MS based proteomic analysis

SUMMARY:
Blood samples will be tested to identify circulating tumor DNA and plasma protein levels to potentially improve prediction of long term prognosis and guide treatment options of patients with hepatocellular carcinoma underwent surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first diagnosis of HCC.
* Patients with HCC who are to undergo surgical treatment, with or without neoadjuvant therapy.
* Ability to obtain tissue sample for ctDNA analysis and detectable baseline ctDNA level.

Exclusion Criteria:

* Patients with secondary liver cancer, or intrahepatic cholangiocarcinoma.
* Any other concurrent malignancy.
* History of organ transplant or hepatic encephalopathy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll male and female subjects with HCC treated with definitive surgery,with or without neoadjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Correlation between ctDNA level and recurrence-free survival (RFS) | 1 years
  ctDNA measurements will be made at baseline and 1 months, 3 months, 6 months, 12 months after surgery. RFS will be assessed by standard radiographic imaging.
Correlation between specific plasma protein expression level and recurrence-free survival (RFS) | 1 years
  plasma proteomic measurements will be made at baseline and 1 months, 3 months, 6 months, 12 months after surgery. RFS will be assessed by standard radiographic imaging.

SECONDARY OUTCOMES:
Correlation between tumor mutation numbers and recurrence-free survival (RFS) | 1 years
  Patients with available tumor tissues were sequenced to identify their specific tumor variants.The correlation of mutation numbers and RFS will be analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No